CLINICAL TRIAL: NCT06861595
Title: USING THE ACCUVEIN DEVICE FOR PATIENTS WHO ARE DIFFICULT TO PERFUSE
Acronym: VAV-AV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/0357/HP
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Patient Who Are Difficult to Infuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- accuvein (Experimental)
  Interventions: Device: accuvein
- with out accuvein (Other)
  Interventions: Other: with out accuvein

INTERVENTIONS:
Device: accuvein — intravenous route with accuvein
  Arms: accuvein
Other: with out accuvein — intravenous route with out accuvein
  Arms: with out accuvein

SUMMARY:
Prior to any examination related to the clinical investigation, the investigator (IDE) will check the eligibility criteria of the person undergoing the research, and will inform and obtain the free, informed and written consent of the person undergoing the research.

The patient will then be randomised into one of two groups (insertion of a intravenous route with the AccuVein device vs. insertion of a VVP without the AccuVein device). After randomisation, the TEC or qualified person starts the stopwatch as soon as the tourniquet is applied.

The nurse makes a first attempt to perfuse the patient. The TEC or the qualified person will stop the stopwatch when the nurse checks the patency of the first attempt at perfusion and signals its success, or when the nurse withdraws the needle if the first attempt is unsuccessful. The pain felt by the patient will be assessed by the nurse using the self-assessment scale from 0 to 10 at the end of the first attempt.

If the first attempt at VVP insertion fails, the choice of conditions and personnel involved in carrying out further attempts will be left to the discretion of the nurse.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients who are difficult to infuse according to the nurse's subjective assessment after the tourniquet has been applied; this may particularly concern patients who are obese, dark-skinned, multi-drug users, sickle-cell anaemia sufferers, drug addicts, elderly with fragile skin and subcutaneous haematomas
* Patients with a medical prescription for intravenous route
* Patients affiliated to a social security scheme
* For women of childbearing age: effective contraception (oral contraceptives, intra-uterine devices or condoms) or post-menopausal women (no menstrual period for 12 months).
* Patient has read and understood the information letter and signed the consent form

Exclusion Criteria:

* Contraindication to fitting a intravenous route (burns to all four limbs, etc.)
* Extreme urgency to have a intravenous route, incompatible with the study, because of a loss of chance due to loss of time
* Patients unable to consent to participation in research
* Pregnant or breastfeeding women or women in labour
* Person deprived of liberty by administrative or judicial decision or person placed under court protection/guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Successful first attempt at intravenous route insertion defined by a functional perfusion placed in a vein | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No